CLINICAL TRIAL: NCT02431819
Title: Single Center Prospective Study Evaluating the Safety of Progressive Compressive Stockings for the Treatment of Venous Insufficiency in Patients With Peripheral Arterial Disease
Brief Title: Evaluation of the Safety of Compressive Socks to Treat Venous Insufficiency in Patients With Peripheral Arterial Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1408064
Record Dates: First submitted 2015-04-28; First posted 2015-05-01 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Peripheral Arterial Disease; Venous Insufficiency
Keywords: Peripheral Arterial Disease; Progressive compressive stockings
MeSH Terms: conditions — Peripheral Arterial Disease; Venous Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- contention socks (Experimental): Patients wear evolutive contention socks during 15 days.
  Interventions: Device: contention socks

INTERVENTIONS:
Device: contention socks — Patients wear contention socks during 15 days.

SUMMARY:
Elastic compression stockings are recommended in the treatment venous insufficiency. Degressive compressive stockings have been used for many decades and are characterized by a high pressure applied at the ankle and a decreasing pressure from the ankle to the knee. Progressive compressive stockings were developed to have a maximal pressure at the calf. This concept is based on the calf pump role in the venous return. Patients with PAD (Peripheral Arterial Disease) often suffer from venous insufficiency. But elastic compression stockings are strictly contraindicated for patients with PAD because highest pressures on ankle could slow down the superficial microcirculation.

On patients with PAD and venous insufficiency, the progressive compressive stockings could be well indicated. Strongest pressure at the calf should increase the pump effect and the muscle mechanical efficiency during the walk without deleterious effect.

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering from a PAD (systolic pressure index ≥ 0,60 and ≤ 0,75) and having moderate venous insufficiency or classified as C1s to C4 using the CEAP classification
* Age over 18 years
* French health insurance
* Signed informed consent

Exclusion Criteria:

* Hypertension not controlled or hypertensive crisis (risk of non reproducibility of SPI and TBI)
* Diabetes
* Mediacalcosis (SPI not computable)
* Inflammatory arterial diseases of the lower limb
* Permanent edema, lipedema and lymphedema
* Wound and fragile skin
* Phlegmatia coerulea dolens
* Septic thrombophlebitis
* Severe coronary artery disease
* Oozing and infectious skin diseases, skin ulcers
* Known hypersensitivity to components of the study compressive stockings

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-02; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
the absence of worsening of PAD after 15 days of progressive compressive stockings ware | Day 15
  The primary endpoint is a safety one: the absence of worsening of PAD after 15 days of progressive compressive stockings ware. A worsening is defined as:
  * Worsening of the systolic ankle pressure index (SPI) defined by a relative reduction of the SPI higher than 15% compared to the index value at inclusion,
  * Worsening of the toe-brachial index (TBI) defined by a relative reduction of TBI higher than 15% compared to the index value at inclusion,
  * Relative reduction of the number of active and repetitive ankle extensions in upright position higher than 25% compared to the index value at inclusion.
  If at least one of these criteria is met, the PAD will be considered as worsening. If none of these criteria is met, the patient will be considered as no worsening.

SECONDARY OUTCOMES:
The evolution of the systolic ankle pressure index (SPI) defined by a relative reduction of the SPI higher than 15% compared to the index value at inclusion, | Day 15
The evolution of the toe-brachial index (TBI) defined by a relative reduction of TBI higher than 15% compared to the index value at inclusion, | Day 15
The relative reduction of the number of active and repetitive ankle extensions in upright position higher than 25% compared to the index value at inclusion. | Day 15
Change of the walking distance on treadmill compared to the walking distance at inclusion | Day 15
Peripheral artery disease symptoms: muscle pain after physical effort, aches, cooling sensation, and paresthesia. | Day 15
Venous insufficiency symptoms | Day 15
Leg heaviness and tiredness leg | Day 15
Pain leg evaluated by visual analogic scale | Day 15
Absence of trophic disorder (new wound or ulcer) | Day 15
Progressive compressive stockings compliance | Day 15
  Progressive compressive stockings compliance will be evaluated by the number of patients stopping wearing the compression before day 15 and reasons for stopping. Patient feeling will also be recorded as free text.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick MISMETTI, MD PhD, Principal Investigator — CHU de SAINT-ETIENNE; Serge COUZAN, MD, Study Director — Clinique Mutualiste Chirurgicale
Locations (2):
- France (2):
  - CHU de Saint-Etienne, Saint-Etienne
  - Clinique Mutualiste Chrirugicale, Saint-Etienne